CLINICAL TRIAL: NCT02731625
Title: Effects of a Regimented Kettlebell Training Program Across Measures of Power and Performance: A Randomized Controlled Trial
Brief Title: Kettlebell Training Measured Across Power and Performance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Less enrollment than expected. Would have been grossly underpowered
Sponsor: Keller Army Community Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brian Stoltenberg, Physical Therapist, Keller Army Community Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16-011
Record Dates: First submitted 2016-03-19; First posted 2016-04-07 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Athletic Performance; Weight Lifting
Keywords: Kettlebell training; High-intensity interval training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kettlebell Training (Experimental): Army Physical Readiness Training (PRT) with kettlebell training in place of strength training circuits
  Interventions: Other: Kettlebell training; Other: Army Physical Readiness Training
- Army Physical Readiness Training (Active Comparator): Army Physical Readiness Training (PRT) per Army Field Manual 7-22
  Interventions: Other: Army Physical Readiness Training

INTERVENTIONS:
Other: Kettlebell training — Kettlebell training will be performed in 30 second work:rest intervals. Total training time will progress from 10 minutes at the beginning of the study to 20 minutes at the end.
  Arms: Kettlebell Training
Other: Army Physical Readiness Training — Army Physical Readiness Training per Army Field Manual 7-22

SUMMARY:
The purpose of this study is to investigate the performance benefits of supplementing Army standard Physical Readiness Training (PRT) with a defined kettlebell (KB) deadlift and swing training program as compared to standalone PRT. Power and performance will be measured on horizontal (broad) and vertical jumps, 40 yard sprint, 60 yard shuttle, and the Army Physical Fitness Test (APFT). It is hypothesized that the unique force distributions of kettlebell training will promote improved power, particularly across the horizontal plane, when compared to standalone Army PRT. Findings will potentially provide insight as to how Army units can effectively utilize kettlebells to further diversify their training programs.

DETAILED DESCRIPTION:
A sample of 140 subjects will be recruited from the remedial physical training population of the Corps of Cadets. This will be achieved through regular communication with company level Tactical Officers (TAC) and Physical Development Officers (PDO). Upon consent, unit integrity will be maintained as the teams of Cadets will be randomized to either the Army standard PRT group or the KB group. Once groups are assigned, PDO's will be provided with their training calendars for the upcoming eight week period and a kettlebell safety/familiarization session will be arranged for all units in the KB group.

Prior to the start of training, all subjects will undergo a pre-assessment on the following performance measures: broad jump, vertical jump, 40 yard sprint and 60 yard shuttle. Current APFT scores will be collected from the West Point Academy Management System (AMS). After the assessment, those assigned to the PRT group will conduct training in accordance with Army Field Manual 7-22 (sustainment phase activity). The KB group will conduct the same training with the exception of kettlebell exercise in place of strength training circuits (this occurs on alternating days). KB exercise will initially be instructed by the principal investigator (certified kettlebell instructor through Crossfit®), but once independence with exercise is noted, the principal investigator's role will become supervisory and continued KB exercise will be executed under the leadership of unit PDO's. Upon conclusion of the eight week training program, all subjects will undergo a post-assessment consisting of the same measures noted previously. Follow on APFT scores will be collected either from West Point AMS for graded tests or from the TACs/PDOs for diagnostic tests.

Once data collection is complete, analysis will be performed using SPSS version 19. A 2x2 mixed-model analysis of variance will be performed with application of Sidak's multiple comparison test to determine if statistical significance has been reached.

ELIGIBILITY:
Inclusion

* Male and Female Cadets
* Age 18-27
* Emancipated minor at age 17
* Remedial physical training participant

Exclusion

* Self-reported pregnancy
* Participants who are not fluent in English
* History of a musculoskeletal injury in the last month
* Any history of a spondylolisthesis
* History of an orthopedic surgery in the last six months
* Condition that results in surgery during the study,
* Missing >1 exercise session per week

Ages: 17 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in Horizontal (Broad) Jump at 8 weeks | Baseline and 8 week re-assess
  This test will be used to assess leg strength and power. Subjects will be advised to assume a standing position with toes directly behind a taped start line. On their own command, subjects will jump as far as they can along a tape measure secured to the floor. Subjects will be encouraged to bend at the knees and hips and swing their arms to assist the jump. Subjects must jump from both feet and land with both feet without falling backward. The distance jumped will be recorded to the nearest centimeter, from the start line to the point of closest heel contact. Subjects will be given three attempts at this test
Change in 40 Yard Sprint at 8 weeks | Baseline and 8 week re-assess
  This test will be used to assess anaerobic power and speed. Subjects will be advised to assume a three-point position behind a start line. On their own command, subjects will run as fast as they can through the finish line. Time will stop when they cross the timing gate. Subjects will be given a single attempt at this test.

SECONDARY OUTCOMES:
Change in Vertical Jump at 8 weeks | Baseline and 8 week re-assess
  This test will be used to assess leg strength and power. Subjects will first be advised to assume a standing position with their feet together and legs straight, positioned directly beneath the measuring device. Without jumping, subjects will reach one arm upward, touching the highest vane they can. This will be recorded as standing reach. Subjects will then be advised to assume a standing position with feet shoulder width apart, again positioned directly beneath the measuring device. Subjects will then, on their own command, jump straight up as high as they can, striking the highest vane they can reach with one hand. Subjects will be encouraged to bend at the knees and hips and swing their arms to assist the jump. Subjects must jump from both feet and land with both feet below the measuring device. Subjects will be given three attempts at this test.
Change in 60 Yard Shuttle at 8 weeks | Baseline and 8 week re-assess
  This test will be used to assess speed and agility. This test is designed as a basic out-and-back shuttle run and one hand must touch each mark as a subject changes directions. Subjects will be advised to assume a three-point position behind the start line. On their own command, subjects will run out to the 5 yard line then return back to the start. Without pause, this pattern will be repeated for the 10 and the 15 yard lines. Time will begin upon subjects initial movement out of the start and will end upon crossing the finish line. Subjects will be given a single attempt at this test.

OTHER OUTCOMES:
Change in Army Physical Fitness Test at 12 weeks | Baseline and up to 12 weeks
  This study will not administer any fitness tests; scores will be pulled from established databases of tests already scheduled as part of cadet requirements.

CONTACTS AND LOCATIONS:
Locations (1):
- Arvin Cadet Physical Development Center, Physical Therapy Clinic, West Point, New York, United States

IPD SHARING:
Plan to Share IPD: No